CLINICAL TRIAL: NCT00680069
Title: A Randomized, Double-Blinded, Phase I/II Study of the Safety, Reactogenicity, and Immunogenicity of an Inactivated Influenza Vaccine Derived From A/H5N1/Indonesia/05/05 (Clade 2) in Healthy Adults and Elderly Who Participated in a Previous A/H5N1/Vietnam/1203/2004 (Clade 1) Vaccine Study
Brief Title: H5N1 (Clade 2) Vaccination of Adults and Elderly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-0022
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2015-08

CONDITIONS: Influenza
Keywords: avian influenza,H5N1,Influenza,parent protocol
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- High Dose Group (Experimental): Volunteers will receive 90 mcg IM. Subjects who received previous clade 1 vaccine will get 1 dose, clade 1 vaccine-naive subjects receive 2 doses 28 days apart
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005
- Low Dose Group (Experimental): Volunteers will receive 15 mcg intramuscularly (IM). Subjects who received previous clade 1 vaccine will get 1 dose, clade 1 vaccine-naive subjects receive 2 doses 28 days apart.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005 — Inactivated monovalent subvirion influenza A/H5N1/Indonesia/05/05 (clade 2) vaccine administered via intramuscular injection. Low Dose Group will receive 15 mcg intramuscularly (IM), High Dose Group will receive 90 mcg IM. Subjects who received previous clade 1 vaccine will receive 1 dose, clade 1 vaccine-naive subjects will receive 2 doses 28 days apart.

SUMMARY:
The purpose of this research study is to study the safety and effectiveness of vaccinating individuals who have previously received an avian influenza vaccine derived from one type of H5N1 virus with a vaccine derived from a different type of avian influenza virus. A second reason for this study is to compare responses in people who have received two different but similar types of H5N1 vaccine to the responses in subjects who receive 2 doses of only the H5N1 vaccine used in this study. The information obtained may provide important information into the usefulness of a pre-pandemic vaccination. Participants will include 600 healthy adult volunteers, ages 19 and older, in the United States. Study procedures include: physical exams, vaccination with either a low dose (15 micrograms) or high dose (90 micrograms) of vaccine, blood samples, and maintaining a memory aid to record oral temperatures and side effects. Study participation will be approximately 7 months.

DETAILED DESCRIPTION:
The goals of this study are to investigate the safety, reactogenicity, and immunogenicity of a single dose of monovalent subvirion influenza vaccine produced from a clade 2 A/H5N1 vaccine administered by intramuscular injection to healthy adults and the elderly who have previously received at least 2 doses of clade 1 A/H5N1 vaccine. In addition, this study will compare these results to individuals who are receiving 2 doses of the clade 2 A/H5N1 vaccine for the first time. The primary objective of the study is to compare the immune response following a single low-dose (15 mcg) to a single high-dose (90 mcg) of influenza vaccine derived from the clade 2 virus A/H5N1/Indonesia/05/05 in individuals who have previously received at least 2 doses of an influenza vaccine derived from the clade 1 virus A/H5N1/Vietnam/1203/2004 (A/VN/1203/04). The secondary objectives will: compare the immune response following a single low-dose (15 mcg) or single high-dose (90 mcg) of influenza vaccine derived from the clade 2 virus A/H5N1/Indonesia/05/05 in individuals who have previously received at least 2 doses of an influenza vaccine derived from the clade 1 virus A/H5N1/Vietnam/1203/2004 (A/VN/1203/04) to a group that has not received any previous A/H5N1 vaccine but who will receive 2 doses of an influenza vaccine derived from the clade 2 virus A/H5N1/Indonesia/05/05; evaluate the factors associated with immunologic response to a single dose of a vaccine derived from a clade 2 virus among individuals who have previously received at least 2 doses of vaccine derived from a clade 1 virus; evaluate the safety of a single dose of subvirion inactivated vaccine derived from the clade 2 virus A/H5N1/Indonesia/05/05 in individuals who have previously received at least 2 doses of an influenza vaccine derived from the clade 1 virus A/H5N1/Vietnam/1203/2004 (A/VN/1203/04); explore immunologic responses following vaccination with a clade 2 vaccine from A/H5N1/Indonesia/05/05 to influenza strains other than A/H5N1/Indonesia/05/05, including A/VN/1203/04; evaluate the immune responses of previously unvaccinated individuals after 1 or 2 doses of clade 2 virus A/H5N1/Indonesia/05/05 vaccine; and evaluate the duration of antibody responses following 1 or 2 doses of vaccine derived from the clade 2 virus A/H5N1/Indonesia/05/05. This study will recruit 600 healthy volunteers aged 19 years or older, in the United States, who have previously participated in a linked DMID-sponsored study. This study is linked to DMID protocols 04-063, 05-0090, 04-076, 05-0015, 05-0127, 05-0141, 06-0089, 04-062, 06-0052, and 08-0030. The study will be conducted at up to 7 vaccine centers. Subjects who previously received at least 2 doses of the clade 1 vaccine derived from the A/H5N1/Vietnam/1203/2004 virus will be randomized to receive a single dose of either 15 mcg or 90 mcg of a clade 2 vaccine derived from the A/H5N1/Indonesia/05/05 virus in a 1:1 ratio. H5 naïve subjects who previously received at least 2 doses of a placebo will be randomized to receive 2 doses of either the 15 mcg or 90 mcg of a clade 2 vaccine derived from the A/H5N1/Indonesia/05/05 virus in a 1:1 ratio. Volunteers will be observed in the clinic for 15 minutes after inoculation, and will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 8 days following each vaccination. Volunteers will be contacted by telephone 1 to 3 days after each vaccination to assess for the occurrence of AEs, and they will return to the clinic 8-10 days after each vaccination for AE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the memory aid. T

ELIGIBILITY:
Inclusion Criteria:

-The subject must have previously received at least 2 doses via the intramuscular route of placebo or vaccine derived from A/H5N1/VN/1203/04 as part of one of the following DMID Protocol Nos.: 04-062, 04-063 (and 05-0090), 04-076, 05-0015, 05-0127, 05-0141, or 06-0089; or the subject must have received placebo intramuscularly as part of DMID Protocol No. 06-0052. -The subject must be 19 years old or older. -Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception, including, but not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices), during the study period between enrollment and 30 days following receipt of the last dose of vaccine. -For a female subject of childbearing potential, she must have a negative pregnancy test (urine or serum) within 24 hours prior to vaccination. -The subject is in good health, as determined by vital signs (heart rate less than 100 bpm; blood pressure: systolic greater than or equal to 90 mm Hg and less than or equal to 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature less than 100.0 degrees Fahrenheit), medical history to ensure stable medical condition, and a targeted physical examination, when necessary, based on medical history. A systolic blood pressure of less than or equal to 160 and a diastolic blood pressure of less than or equal to 90 is acceptable in subjects greater than 65 years of age. -The subject is able to understand and comply with the planned study procedures, including being available for all study visits. -The subject has provided informed consent prior to any study procedures.

Exclusion Criteria:

-The subject is allergic to eggs, egg products, chicken or egg proteins or other components of the vaccine (including gelatin, formaldehyde, octoxinol and thimerosal). -The subject is a woman who is breastfeeding or intends to become pregnant during the study period between enrollment and 30 days following receipt of the last dose of vaccine. -The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months. -The subject has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. An active neoplastic disease is defined as treatment for neoplastic disease within the past 5 years. -The subject has long-term (greater than 2 weeks) use of oral or parenteral glucocorticoids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed). -The subject received immunoglobulin or another blood product within the 3 months prior to enrollment in this study. -The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days (or 56 days for prior placebo recipients). -The subject has an acute or chronic medical condition that would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to: solicited reactogenicity symptoms, history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long as there has been no dose adjustment with the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Association Functional Class III or IV); an arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries or transient ischemic attack). -The subject has a history of a severe reaction following receipt of an influenza virus vaccine. -The subject has an acute illness or an oral temperature greater than 99.9 degrees Fahrenheit (37.7 degrees Celsius) within 3 days prior to enrollment or vaccination. -The subject is currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study. -The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol. -The subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis. -The subject has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others. -The subject is receiving psychiatric drugs. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study. -The subject has a history of alcohol or drug abuse in the 5 years prior to enrollment. -The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection. -The subject has a history of Guillain-Barré syndrome. -The subject has any condition that the investigator believes may interfere with successful completion of the study. The subject plans to enroll in another clinical trial that has a study intervention such as a drug, biologic, or device that could interfere with safety assessment of the investigational product at any time during the study period.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Immune responses approximately 28 days after one dose of an H5N1 clade 2 vaccine. | Approximately Day 28.

SECONDARY OUTCOMES:
Immunologic outcomes include antibodies generated against strains other than A/Indonesia/05/05. | Blood samples taken prior to vaccination on Day 0, and 28 days and 6 months after receipt of last vaccination testing.
Safety outcomes include frequencies and severities of adverse events (AEs) in the high- and low-dose groups in aggregate, and in other strata previously identified. | Duration of Study

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Result] Winokur PL, Patel SM, Brady R, Chen WH, El-Kamary SS, Edwards K, Creech CB, Frey S, Keitel WA, Belshe R, Walter E, Bellamy A, Hill H. Safety and Immunogenicity of a Single Low Dose or High Dose of Clade 2 Influenza A(H5N1) Inactivated Vaccine in Adults Previously Primed With Clade 1 Influenza A(H5N1) Vaccine. J Infect Dis. 2015 Aug 15;212(4):525-30. doi: 10.1093/infdis/jiv087. Epub 2015 Feb 23. PMID 25712967
- [Derived] Belshe RB, Frey SE, Graham IL, Anderson EL, Jackson LA, Spearman P, Edupuganti S, Mulligan MJ, Rouphael N, Winokur P, Dolor RJ, Woods CW, Walter EB, Chen WH, Turley C, Edwards KM, Creech CB, Hill H, Bellamy AR; National Institute of Allergy and Infectious Diseases-Funded Vaccine and Treatment Evaluation Units. Immunogenicity of avian influenza A/Anhui/01/2005(H5N1) vaccine with MF59 adjuvant: a randomized clinical trial. JAMA. 2014 Oct 8;312(14):1420-8. doi: 10.1001/jama.2014.12609. PMID 25291578